CLINICAL TRIAL: NCT01233076
Title: Clinical Comparison of Two Daily Disposable Contact Lenses in a Population of Daily Disposable Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-337-C-034
Record Dates: First submitted 2010-11-01; First posted 2010-11-03 (Estimated); Results first posted 2011-09-08 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

ARMS (2):
- Nelfilcon A / Narafilcon B (Other): Nelfilcon A worn first, with narafilcon B worn second. Each product worn bilaterally in a daily wear, daily disposable basis for one week.
  Interventions: Device: Nelfilcon A contact lens; Device: Narafilcon B contact lens
- Narafilcon B / Nelfilcon A (Other): Narafilcon B worn first, with nelfilcon A worn second. Each product worn bilaterally in a daily wear, daily disposable basis for one week.
  Interventions: Device: Nelfilcon A contact lens; Device: Narafilcon B contact lens

INTERVENTIONS:
Device: Nelfilcon A contact lens — Commercially marketed, spherical contact lens for daily wear, daily disposable use
  Other Names: DAILIES AquaComfort Plus
Device: Narafilcon B contact lens — Commercially marketed (US), spherical contact lens for daily wear, daily disposable use
  Other Names: 1-DAY ACUVUE TruEye

SUMMARY:
The purpose of this study is to evaluate the performance of two commercially marketed daily disposable contact lenses in a population of daily disposable contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Currently wearing daily disposable lenses in daily wear, daily disposable modality, except DAILIES AquaComfort Plus and 1-DAY ACUVUE TruEye.
* Able to wear study lenses in the available powers from -1.00D to -6.00D.
* Other protocol-defined inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Eye injury within twelve weeks of enrollment.
* History of corneal or refractive surgery.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Currently enrolled in any clinical trial.
* Currently wearing DAILIES AquaComfort Plus or 1-DAY ACUVUE TruEye lenses.
* Monovision correction during the study.
* Other protocol-defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This reporting group includes all enrolled and dispensed participants.
Period: Period 1, One Week
Arm/Group | Nelfilcon A / Narafilcon B | Narafilcon B / Nelfilcon A
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0
Period: Period 2, One Week
Arm/Group | Nelfilcon A / Narafilcon B | Narafilcon B / Nelfilcon A
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all enrolled and dispensed participants.
Arm/Group | Overall
Number analyzed (Participants) | 60
Age Continuous [Mean (Standard Deviation); unit: years] | 30.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Vision Quality
Description: Overall vision quality, as interpreted by the participant and recorded on a questionnaire as a single, retrospective evaluation of 1 week of wear. Overall vision quality is evaluated binocularly and rated on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 1 week of wear
Population: Analysis conducted per protocol, with exclusions due to reasons such as: major protocol deviations as determined by masked review; discontinuations; and/or missing responses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Nelfilcon A: Commercially marketed, spherical contact lenses worn bilaterally in a daily wear, daily disposable manner for one week.
- Narafilcon B: Commercially marketed (US), spherical contact lenses worn bilaterally in a daily wear, daily disposable manner for one week.
Arm/Group | Nelfilcon A | Narafilcon B
Number analyzed (Participants) | 59 | 59
units on a scale | 8.2 (1.7) | 8.7 (1.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial: 41 days.
Description: This reporting group includes all enrolled and exposed subjects.
Arm/Group | Nelfilcon A | Narafilcon B
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.